CLINICAL TRIAL: NCT07230756
Title: A Prospective Cohort Study of Coronary Heart Disease Complicated With Ischemic Mitral Regurgitation in China
Brief Title: Coronary Heart Disease Complicated With Ischemic Mitral Regurgitation in China
Acronym: China-IMR
Status: Not yet recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2024-GSP-TJ-7
Record Dates: First submitted 2025-01-02; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-12

CONDITIONS: Ischemic Mitral Regurgitation; Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Investigators will collect blood samples from up to 2,500 patients, separate patients' plasma, serum, and peripheral blood RNA, and store them long-term in the biobank of the National Center for Cardiovascular Diseases. These samples will be used for future extended studies, such as nested cohort studies , with the aim of discovering new biomarkers and other purposes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- GDMT Group
- Non-GDMT Group

SUMMARY:
This project will rely on the established multi-center cooperation platform for total valve disease and based on the Carpentier classification, which is newly proposed and widely recognized by the academic community, and will specifically target the population with coronary heart disease combined with Ischemic Mitral Regurgitation（IMR） to conduct a nationwide, multi-center, single valve disease, prospective cohort. Research. From November 2025 to December 2025, 6,000 patients with coronary heart disease combined with moderate or above IMR were consecutively selected from outpatients or inpatients in 21 regional medical centers across the country, and clinical characteristics, imaging data, and serology were collected. Information, drug/surgical intervention status and clinical outcome indicators were included in the clinical follow-up at baseline, 3 months, 6 months, 12 months and 24 months respectively. The main research objectives are to describe the disease characteristics, treatment status and clinical outcomes of coronary heart disease patients with IMR; to evaluate the current application status of GDMT strategies in IMR diagnosis and treatment practice and its impact on mid- and long-term prognosis. The secondary research objectives are to identify factors affecting prognosis, construct a risk stratification model for mid- and long-term prognosis, and discover new molecular markers.

This project will for the first time construct the world's largest clearly defined cohort of coronary heart disease combined with IMR. Its research results can provide high-quality data and decision-making basis for precise diagnosis and treatment of IMR populations. Therefore, this project has important scientific research value and clinical guidance significance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, secondary mitral regurgitation discovered during outpatient visit or hospitalization;
* Have definite coronary heart disease
* Cardiac ultrasound: consistent with mitral regurgitation caused by myocardial ischemia or myocardial infarction:

  1. Segmental wall motion abnormality or
  2. Mitral regurgitation is consistent with Carpentier type IIIb (eccentric regurgitation)
* Cardiac ultrasound prompts: moderate or above ischemic mitral regurgitation

Exclusion Criteria:

* Patients within the past year or currently participating in other clinical studies;
* Primary mitral regurgitation (such as mitral valve prolapse, perforation, chordae tendineae rupture, etc.);
* Dilated cardiomyopathy, hypertrophic cardiomyopathy and other diseases;
* Moderate and above aortic stenosis/regurgitation, mitral stenosis, tricuspid stenosis, etc.;
* Patients who have undergone cardiac valve intervention/surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with coronary heart disease combined with ischemic mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of heart failure hospitalization and all-cause death | 3, 6, 12, 24 months
  Time to first occurrence of either hospitalization for heart failure or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Change in mitral regurgitation severity | 3 month, 6 month, 12 month, 24 month
  Change in mitral regurgitation (MR) grade from baseline to 24 months as assessed by echocardiography, measured using standard semiquantitative grading (none, mild, moderate, severe).
All-cause mortality | 3 month, 6 month, 12 month, 24 month
  Incidence of death due to any cause during the follow-up period
Hospitalization for heart failure | 3, 6, 12, 24 months
  Incidence of unplanned hospital admission primarily for management of heart failure symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Erli Zhang, MD, PhD, Principal Investigator — China National Center for Cardiovascular Diseases

IPD SHARING:
Plan to Share IPD: No